CLINICAL TRIAL: NCT00751907
Title: Impact of Atorvastatin on Cerebral Perfusion and Endothelial Function
Brief Title: Cerebral and Peripheral Perfusion Pilot Study
Acronym: CAPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IA0138; K23AG026752 (NIH); Pilot Award (Other Grant/Funding Number: Wisconsin Comprehensive Memory Program Pilot Award)
Record Dates: First submitted 2008-09-10; First posted 2008-09-12 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer's Disease
Keywords: Cerebral blood flow
MeSH Terms: conditions — Alzheimer Disease | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): 40mg Atorvastatin nightly for 4 months
  Interventions: Drug: atorvastatin
- Placebo (Placebo Comparator): matching placebo nightly for 4 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: atorvastatin — 40mg daily for 4 months
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Placebo — Matching placebo daily for 4 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the hypothesis that in middle-aged, asymptomatic, adult children of persons with Alzheimer's disease (AD), atorvastatin therapy will beneficially affect mechanisms thought to contribute to AD risk by improving blood flow in the brain, improving cerebral perfusion, increasing brain activity patterns, and improving blood vessel function.

DETAILED DESCRIPTION:
Treatment with cholesterol-lowering medications, specifically statins, is associated with up to a 73% reduction in the prevalence of AD, suggesting a potentially promising role for statins in the prevention of AD. In order to better understand the mechanisms through which statins may possibly modify blood AD risk, this study evaluated whether administration of atorvastatin favorably altered blood flow in the brain (measured by magnetic resonance imaging (MRI)) and blood vessel function (measured by ultrasound).

Participants attended 3 visits over the course of the 4-month study. At the initial visit, participants completed a short questionnaire about their past medical history and medication history. At the baseline visit, participants were randomized in a 1:1 ratio to receive atorvastatin 40 mg nightly vs. matching placebo. At baseline and follow-up visits, participants provided an update on medical problems and medications, reviewed any potential side effects, and had fasting blood tests collected for safety monitoring, including liver and muscle enzyme monitoring. In addition, all participants had MRI and ultrasound measures collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult (ages 40-65) children of parent with documented Alzheimer's disease

Exclusion Criteria:

* Current use of cholesterol lowering medication
* History of liver disease
* History of adverse reaction to statin medications
* Elevated lab values (CK and creatinine)
* Use of medications that counteract with atorvastatin
* History of dementia
* Currently pregnant
* Use of large quantities of grapefruit juice (more than 1 quart/day)
* Current involvement in another investigational drug study
* Contraindications to MRI

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change in regional cerebral blood flow (rCBF) | Baseline and 4 months
  rCBF , a measure of cerebral perfusion, is the primary outcome. rCBF was measured by arterial spin-labeling magnetic resonance imaging and used to evaluate effects of atorvastatin vs placebo

SECONDARY OUTCOMES:
Change in Endothelial function | Baseline and 4 months
  Brachial artery reactivity was used to measure endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M. Carlsson, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Karen Lazar, Madison, Wisconsin, United States

REFERENCES:
- [Background] Newman GC, Delucia-Deranja E, Tudorica A, Hospod FE, Patlak CS. Cerebral blood volume measurements by T*2-weighted MRI and contrast infusion. Magn Reson Med. 2003 Oct;50(4):844-55. doi: 10.1002/mrm.10591. PMID 14523972
- [Background] Sorensen KE, Celermajer DS, Spiegelhalter DJ, Georgakopoulos D, Robinson J, Thomas O, Deanfield JE. Non-invasive measurement of human endothelium dependent arterial responses: accuracy and reproducibility. Br Heart J. 1995 Sep;74(3):247-53. doi: 10.1136/hrt.74.3.247. PMID 7547018
- [Background] Wassmann S, Ribaudo N, Faul A, Laufs U, Bohm M, Nickenig G. Effect of atorvastatin 80 mg on endothelial cell function (forearm blood flow) in patients with pretreatment serum low-density lipoprotein cholesterol levels <130 mg/dl. Am J Cardiol. 2004 Jan 1;93(1):84-8. doi: 10.1016/j.amjcard.2003.09.018. PMID 14697473
- [Background] Stein JH, Keevil JG, Wiebe DA, Aeschlimann S, Folts JD. Purple grape juice improves endothelial function and reduces the susceptibility of LDL cholesterol to oxidation in patients with coronary artery disease. Circulation. 1999 Sep 7;100(10):1050-5. doi: 10.1161/01.cir.100.10.1050. PMID 10477529
- [Background] Sever PS, Dahlof B, Poulter NR, Wedel H, Beevers G, Caulfield M, Collins R, Kjeldsen SE, Kristinsson A, McInnes GT, Mehlsen J, Nieminen M, O'Brien E, Ostergren J; ASCOT investigators. Prevention of coronary and stroke events with atorvastatin in hypertensive patients who have average or lower-than-average cholesterol concentrations, in the Anglo-Scandinavian Cardiac Outcomes Trial--Lipid Lowering Arm (ASCOT-LLA): a multicentre randomised controlled trial. Lancet. 2003 Apr 5;361(9364):1149-58. doi: 10.1016/S0140-6736(03)12948-0. PMID 12686036
- [Result] Carlsson CM, Xu G, Wen Z, Barnet JH, Blazel HM, Chappell RJ, Stein JH, Asthana S, Sager MA, Alsop DC, Rowley HA, Fain SB, Johnson SC. Effects of atorvastatin on cerebral blood flow in middle-aged adults at risk for Alzheimer's disease: a pilot study. Curr Alzheimer Res. 2012 Oct;9(8):990-7. doi: 10.2174/156720512803251075. PMID 22175654
- See also: Wisconsin Alzheimer's Disease Research Center — http://adrc.wisc.edu/